CLINICAL TRIAL: NCT02519153
Title: Role of Phosphodiesterase 5 Inhibitors (PDE5i) (Sildenafil) in Management of Distal Ureteral Stone
Brief Title: Phosphodiesterase 5 Inhibitors (PDE5i) (Sildenafil) as Medical Expulsive Therapy in Distal Ureteral Stones
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, mohamed awad tharwat, Urology & Nephrology Center, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MThar87
Record Dates: First submitted 2015-06-30; First posted 2015-08-10 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Ureteral Stone; Urolithiasis
Keywords: Phosphodiesterase 5 Inhibitors; PDE5i; Sildinafil
MeSH Terms: conditions — Ureterolithiasis; Urolithiasis | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (Placebo Comparator): patient receive placebo for 4 weeks and followed for passage of stone distal ureter
  Interventions: Drug: Sildenafil
- sildenafil (Active Comparator): patient receive sildenafil 50 mg for 4 weeks once per day and followed for passage of stone distal ureter
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — placebo will take nitrofuratoin once daily for 4 weeks . sildenafil arm will take sildenafil 50 mg once daily for 4 weeks

SUMMARY:
Urolithiasis is one of the most common urological diseases. The risk of urolithiasis is estimated to be between 5% and 12% all over the world with increased incidence in male rather than female (2:1) respectively . Ureteral stones account for 20% from all urinary tract stones, more than 70% of the ureteral stones found in the lower third of the ureter . The incidence of urinary stones has been increasing day by day. Medical expulsive therapy (MET) of ureteral stones is the investigators' concern in this study. Stone location, size, number, ureteral spasm, mucosal edema or inflammation and ureteral anatomy are the factors affecting passage of the ureteral stones. So, MET is based on mechanism that stone passage is facilitated by the relaxation of ureteral smooth muscle , increasing hydrostatic pressure proximal to the stone and decreasing exciting edema . There are many oral medication could be used as MET such as adrenergic blockers, calcium channel blockers, prostaglandin synthesis inhibitors, glyceryl trinitrate and steroid treatment . Calcium-channel blockers and adrenergic α-antagonists are the main that has been proposed to enhance stone passage as expulsive medical therapy. Cyclic nucleotides are degraded by phosphodiesterases enzymes (PDEs). So using of PDE inhibtors may play role in relaxation of smooth muscle of the ureter. A study was done for evaluation of three PDE5 inhibtors, sildenafil , vardenafil and tadalafil, they found that PDE5 inhibitors can reverse the tension of isolated human ureteral smooth muscle via cGMP-mediated pathways.

ELIGIBILITY:
Inclusion Criteria:

1. Male Patient aged from 18-65 years.
2. Lower third ureteric stones at or below sacro-iliac joint .
3. Stone size rang from 5- 10 mm.
4. Unilateral ureteric stone

Exclusion Criteria:

1. Patients who had recurrent fever.
2. Patient underwent ESWL.
3. Patient with rising serum creatinine > 2mg/dl.
4. Patient with history of uretero-vesical reimplantation.
5. Stone larger than 10 mm

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
the percentage of passage of lower ureteric stones. | one year

SECONDARY OUTCOMES:
number of patient need for analgesic treatment during their medical expulsive tharpy | one year